CLINICAL TRIAL: NCT00903760
Title: A Randomized Study of Decitabine Alternating With Clofarabine Versus Decitabine Until Failure in Patients With Higher Risk Myelodysplastic Syndromes (MDS)
Brief Title: Decitabine and Clofarabine in Higher Risk Myelodysplastic Syndromes (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0092; NCI-2011-00263 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; MDS; Leukemia; Decitabine; clofarabine; Dacogen®; Clolar®
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia | interventions — Decitabine; Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decitabine + Clofarabine (Experimental): Drug delivery intravenously (IV) in alternating series of cycles (Decitabine 20 mg/m^2 for 5 days first 3 cycles, then Clofarabine 10 mg/m^2 five days for next 3 cycles), pattern repeats for up to 24 cycles.
  Interventions: Drug: Decitabine; Drug: Clofarabine
- Decitabine (Experimental): Decitabine 20 mg/m^2 IV daily for 5 days for a total of 24 courses.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — Decitabine 20 mg/m^2 by vein daily over 1-2 hours for 5 days for both Group 1 and Group 2. Group 1 receives decitabine on Days 1-5 of Cycles 1-3, 7-9, 13-15, and 19-21; and Group 2 is on Days 1-5 of every cycle.
  Other Names: Dacogen®
Drug: Clofarabine — Clofarabine 10 mg/m^2 by vein daily over 1-2 hours for 5 days on Days 1-5 of Cycles 4-6, 10-12, 16-18, and 22-24.
  Other Names: Clolar®
  Arms: Decitabine + Clofarabine

SUMMARY:
The goal of this clinical research study is to learn if sequential administration of decitabine and clofarabine can help to control MDS better than decitabine alone. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Decitabine is designed to damage cells' DNA (genetic material), which may cause myelodysplastic marrow cells to work more like normal marrow cells.

Clofarabine is designed to interfere with the growth and development of abnormal marrow cells.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups.

* If you are in Group 1, you will receive decitabine and clofarabine.
* If you are in Group 2, you will receive only decitabine.

Study Drug Administration:

Each cycle is 4-8 weeks depending on how you tolerate the drug and how the MDS responds to it.

Group 1:

If you are in Group 1, you will receive the drugs in an alternating series of cycles. This means that you will receive decitabine for the first 3 cycles, then clofarabine for the next 3 cycles, and then repeat. This pattern will continue for up to 24 cycles.

On Days 1-5 of Cycles 1-3, 7-9, 13-15, and 19-21, you will receive decitabine by vein over 1-2 hours.

On Days 1-5 of Cycles 4-6, 10-12, 16-18, and 22-24, you will receive clofarabine by vein over 1-2 hours.

Group 2:

If you are in Group 2, you will receive decitabine by vein over 1-2 hours on Days 1-5 of every cycle.

Study Visits:

On Day 1 of every cycle, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.

Once a week, blood (about 1-2 teaspoons) will be drawn for routine tests.

At the end of Cycle 3, you will have a bone marrow aspirate to check the status of the disease.

If the disease has not gone into remission after Cycle 3, your next bone marrow aspirate will depend on your group. If you are in Group 1, you may have another aspirate about 3 weeks after you begin Cycle 4. After that, you may have an aspirate every 2 weeks (or more often if your doctor feels it is needed) until the response (or lack thereof) is confirmed. If you are in Group 2, you may not have another bone marrow aspirate until after the end of Cycle 6.

You will need to stay in Houston to receive the study drug(s). When you have study visits where you are not receiving study drug(s), these tests can be performed by your local doctor. If your MD Anderson leukemia doctor approves, your study drug can be administered outside MD Anderson by your local doctor.

Length of Study:

You will be on study for up to 24 cycles. You will be taken off study early if the disease gets worse or you experience any intolerable side effects.

Follow-up Visits:

After your last dose of study drug, you will have follow-up visits. You will only have these visits if the disease has responded to the study drug.

* Once a month, blood (about 1 tablespoon) will be drawn routine tests. This can be done at home through your local cancer doctor.
* Every 6 months, you will return to Houston for a physical exam and blood (about 1 tablespoon) will be drawn for routine tests.

This is an investigational study. Clofarabine is FDA approved and commercially available for use in pediatric patients with a type of blood cancer (acute lymphocytic leukemia -- ALL). Its use in patients with MDS is investigational.

Decitabine is FDA approved and commercially available for use in patients with MDS.

Up to 80 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with higher risk MDS (IPSS int-2 or high, or >/= 10% blasts as defined by WHO or FAB). - No prior intensive chemotherapy or high-dose cytarabine (>/= 1 g/m2). - Prior biologic therapies (</= 1 cycle of prior decitabine or azacitidine), targeted therapies, or single agent chemotherapy is allowed. - Off chemotherapy for 2 weeks prior to entering this study with no toxic effects of that therapy, unless there is evidence of rapidly progressive disease. - Hydroxyurea is permitted for control of counts prior to treatment. - Hematopoietic growth factors are allowed. .
2. Age >/= 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
4. Have adequate renal function (serum creatinine </= 1.5 mg/dL)
5. Serum bilirubin </= 1.5 x upper limit of normal (ULN)
6. Aspartate transaminase (AST) or alanine transaminase (ALT) </= 2.5 x ULN
7. Alkaline phosphatase </= 2.5 x ULN
8. Provide signed written informed consent.
9. Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
10. Female patients of childbearing potential must have a negative pregnancy test within 2 weeks prior to enrollment.
11. Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

1. Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
2. Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea. The patient must have recovered from all acute toxicities from any previous therapy.
3. Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment.
4. Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
5. Pregnant or lactating patients.
6. Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
7. Any concurrent malignancy (with the exception of exclusion # 8)
8. Exceptions to inclusion # 7: a) Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed; b) Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: January 28, 2010 to May 7, 2014. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 42 participant enrolled, five were not randomized or treated and are therefore excluded from the trial details. One participant included in group assignment was randomized but not treated as a result of early death.
Period: Overall Study
Arm/Group | Decitabine + Clofarabine | Decitabine
Started | 19 | 18
Completed | 0 (Completed all 24 courses) | 2 (Completed all 24 courses)
Not Completed | 19 | 16
Not completed — Disease Progression/Death | 8 | 6
Not completed — Stem Cell Transplant | 8 | 4
Not completed — Physician Decision | 1 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Off treatment for long period | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decitabine + Clofarabine | Decitabine | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Customized [Number; unit: participants]
  <=29 | 2 | 0 | 2
  30-39 | 0 | 1 | 1
  40-49 | 1 | 0 | 1
  50-59 | 3 | 1 | 4
  60-69 | 4 | 7 | 11
  70-79 | 9 | 8 | 17
  >=80 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 12 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival (EFS) at 1 Year
Description: Percentage of participants with event free survival at 1 year. Event free survival (EFS) where event is defined as either death or transformation to acute myeloid leukemia (AML) (marrow and/or blood blasts >/= 20%)
Time Frame: Assessed at 12 months/1 year
Population: One of 18 participants in the Decitabine arm was not treated due to early death thus is excluded from analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Decitabine + Clofarabine | Decitabine
Number analyzed (Participants) | 19 | 17
percentage of participants | 26 | 65

2. Secondary Outcome: Participant Response
Description: Responses: Complete Remission (CR): Normalization peripheral blood & bone marrow </= 5% bone marrow blasts, no evidence dysplasia; peripheral blood granulocyte >/= 1.0 x 10^9/L, & platelet>/= 100 x 10^9/L. Partial Remission: all CR criteria if abnormal before treatment except marrow blasts decrease =/> 50% compared to pretreatment or a less-advanced MDS disease classification than prior to treatment. Hematologic Improvement: Response maintained 8+ weeks: Hemoglobin (pretreatment < 11 g/dL): improves 1.5 g/dL or reduced by 4 units of red blood cell (RBC) transfusions in 8 weeks compared with pretreatment transfusions in 8 weeks; or Platelet (pretreatment < 100 x 10^9/L): absolute increase >/= 30 x 10^9/L, starting platelet > 20 x 10^9/L OR increase < 20 x 10^9/L to > 20 x 10^9/L and =/> 100%. Neutrophil (pretreatment < 1 x 10^9/L): increase 100% & absolute increase > 0.5 x 10^9/L.
Time Frame: Up to 6 months
Population: One of 18 participants in the Decitabine arm was not treated due to early death thus is excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Decitabine + Clofarabine | Decitabine
Number analyzed (Participants) | 19 | 17
participants
  Complete Remission (CR) | 8 | 9
  Partial Remission (PR) | 0 | 0
  Hematologic Improvement (HI) | 5 | 4

ADVERSE EVENTS:
Time Frame: Adverse event reporting with each course which is repeated every 4 to 8 weeks, up to 4 years.
Arm/Group | Decitabine + Clofarabine | Decitabine
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/18
Other Adverse Events (participants affected / at risk) | 19/19 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine + Clofarabine (N=19) | Decitabine (N=18)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteremia - Escherichia coli (E. coli) (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) — Septic Shock, Bacteremia
Death (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine + Clofarabine (N=19) | Decitabine (N=18)
Urinary tract infection (UTI) (Infections and infestations) | 4 (4) | 5 (5)
Bacteremia -E. Coli (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia-pseudomonas (Infections and infestations) | 1 (1) | 0 (0)
Bilateral joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bilateral lower lobe pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 6 (6)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Deep vein thrombosis -picc line (Vascular disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 9 (9) | 9 (9)
Fracture-femoral neck (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Infection - other (Infections and infestations) | 2 (2) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Left side weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Respiratory infection (Infections and infestations) | 0 (0) | 2 (2)
Lung Infection (Infections and infestations) | 12 (12) | 2 (2)
Muscle weakness in lower limbs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 5 (5) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash-extremities (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vancomycin-resistant enterococci (VRE) (Infections and infestations) | 0 (0) | 1 (1)
sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes